CLINICAL TRIAL: NCT03206749
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled, 3-arm, Parallel-design Study of the Efficacy and Safety of VX-150 for Acute Pain Following Bunionectomy
Brief Title: A Study to Evaluate Efficacy and Safety of VX-150 in Subjects With Acute Pain Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX16-150-103
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VX-150 (Experimental)
  Interventions: Drug: VX-150
- Hydrocodone Bitartrate/Acetaminophen (HB/APAP) (Active Comparator)
  Interventions: Drug: HB/APAP
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-150 — Participants received VX-150 1500 milligram (mg) as first dose, followed by VX-150 750 mg dose every 12 hours (q12h) for 2 days.
  Arms: VX-150
Drug: HB/APAP — Participants received HB 5 mg/APAP 325 mg every 6 hours (q6h) for 2 days.
  Arms: Hydrocodone Bitartrate/Acetaminophen (HB/APAP)
Drug: Placebo — Participants received placebo matched to VX-150 and HB/APAP for 2 days.
  Arms: Placebo

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled, 3-arm, parallel design study to evaluate the efficacy and safety of VX-150 in treating acute pain following bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

Prior to Surgery:

* Body mass index (BMI) of 18.0 to 38.0 kg/m2, inclusive
* Be scheduled to undergo a primary unilateral first metatarsal bunionectomy repair, without collateral procedures, under regional anesthesia (Mayo and popliteal sciatic block) not to include base wedge procedure

After Surgery:

* Subject reported pain of ≥4 on the NPRS, and moderate or severe pain on the Verbal Categorical Rating Scale (VRS) within 9 hours after removal of the popliteal sciatic block on Day 1
* Subject is lucid and able to follow commands
* All analgesic guidelines were followed during and after the bunionectomy

Exclusion Criteria:

Prior to Surgery:

* History in the past 10 years of malignancy, except for squamous cell skin cancer, basal cell skin cancer, and Stage 0 cervical carcinoma in situ
* History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s)
* History of abnormal laboratory results ≥2.5 × upper limit of normal (ULN)
* History of peripheral neuropathy
* A known or clinically suspected infection with human immunodeficiency virus or hepatitis B or C viruses
* Prior medical history of bunionectomy or other foot surgery
* Intolerant of or unwilling to receive hydrocodone, acetaminophen, or ibuprofen
* For female subjects: Pregnant, nursing, or planning to become pregnant during the study or within 90 days after the last study drug dose
* For male subjects: Male subjects with a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 90 days after the last study drug dose

After Surgery:

* Subject had a type 3 deformity requiring a base wedge osteotomy or concomitant surgery such as hammertoe repair; or experienced medical complications during the bunionectomy that, in the opinion of the investigator, should preclude randomization

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Lotus Clinical Research, Pasadena, California
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydrocodone Bitartrate/Acetaminophen (HB/APAP): Participants received HB 5 mg/APAP 325 mg every 6 hours (q6h) for 2 days.
Period: Overall Study
Arm/Group | VX-150 | Hydrocodone Bitartrate/Acetaminophen (HB/APAP) | Placebo
Started | 80 | 81 | 82
Completed | 75 | 78 | 75
Not Completed | 5 | 3 | 7
Not completed — Withdrawal of consent | 5 | 3 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- VX-150: Participants received VX-150 1500 mg as first dose, followed by VX-150 750 mg q12h for 2 days.
- HB/APAP: Participants received HB 5 mg/APAP 325 mg q6h for 2 days.
- Total: Total of all reporting groups
Arm/Group | VX-150 | HB/APAP | Placebo | Total
Number analyzed (Participants) | 80 | 81 | 82 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.87) | 44.8 (13.04) | 45.0 (12.43) | 44.7 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 64 | 65 | 193
  Male | 16 | 17 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 14 | 27 | 62
  Not Hispanic or Latino | 59 | 67 | 55 | 181
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 1 | 0 | 2
  Race: Asian | 8 | 1 | 3 | 12
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Race: Black or African American | 17 | 22 | 17 | 56
  Race: White | 52 | 55 | 59 | 166
  Race: More than one race | 0 | 0 | 1 | 1
  Race: Other | 1 | 2 | 1 | 4
Pain Intensity at Baseline (at 0 hours) as Recorded on Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on scale] — Pain intensity was recorded on 11-point ordinal NPRS, score range: 0 to 10, where 0=no pain and 10=worst imaginable pain.
  units on scale | 6.1 (1.7) | 6.6 (1.6) | 6.1 (1.5) | 6.3 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of the Pain Intensity Difference (SPID) Between VX-150 Versus Placebo as Recorded on a Numeric Pain Rating Scale (NPRS) 0 to 24 Hours After the First Dose
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0 =no pain to 10 =worst possible pain). SPID24 was calculated from 0 to 24 hours and the score range was -240 (worst score) to 240 (best score).
Time Frame: 0 to 24 hours after the first dose
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study drug. As a standard-of-care reference arm, the "HB/APAP" arm was not intended for statistical comparisons to VX-150.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 80 | 82
units on a scale | 36.14 (5.15) | 6.64 (5.03)
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean Difference = 29.50, 95% CI 2-sided [16.61 to 42.40]

2. Secondary Outcome: Time-weighted Sum of the Pain Intensity Difference Between VX-150 Versus Placebo as Recorded on a NPRS 2 to 24 Hours After the First Dose
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0 =no pain to 10 =worst possible pain). SPID22 was calculated from 2 to 24 hours and the score range was -220 (worst score) to 220 (best score).
Time Frame: 2 to 24 hours after the first dose
Population: FAS. As a standard-of-care reference arm, the "HB/APAP" arm was not intended for statistical comparisons to VX-150.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 80 | 82
units on a scale | 34.95 (4.93) | 6.43 (4.82)
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = 28.53, 95% CI 2-sided [16.18 to 40.88]

3. Secondary Outcome: Time-weighted Sum of the Pain Intensity Difference Between VX-150 Versus Placebo as Recorded on a NPRS 0 to 48 Hours After the First Dose
Description: SPID was calculated as the sum of the product of time (in hours) elapsed since previous measurements and pain intensity difference. Pain intensity difference was calculated by subtracting the pain intensity score at given post-dose time points from the baseline pain intensity scores (using pain rating score range: 0 =no pain to 10 =worst possible pain). SPID48 was calculated from 0 to 48 hours and the score range was -480 (worst score) to 480 (best score).
Time Frame: 0 to 48 hours after the first dose
Population: FAS. As a standard-of-care reference arm, the "HB/APAP" arm was not intended for statistical comparisons to VX-150.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 80 | 82
units on a scale | 112.22 (10.57) | 49.43 (10.33)
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = 62.79, 95% CI 2-sided [36.30 to 89.27]

4. Secondary Outcome: Time to Onset of Perceptible Pain Relief After the First Dose of VX-150 Versus Placebo
Description: Time to onset of perceptible pain relief (any pain relief at all after the first dose) reported based on the first stopwatch assessment.
Time Frame: up to 6 hours after the first dose
Population: FAS. As a standard-of-care reference arm, the "HB/APAP" arm was not intended for statistical comparisons to VX-150.
Measure: Median (Full Range); unit: minutes
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 80 | 82
minutes | 26.8 [2 to 177] | 28.3 [5 to 239]
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p = 0.0469, Regression, Cox; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [1.01 to 2.16]

5. Secondary Outcome: Time to Onset of Meaningful Pain Relief After the First Dose of VX-150 Versus Placebo
Description: Time to onset of meaningful pain relief (relief that is meaningful to participants after the first dose) reported based on the second stopwatch assessment.
Time Frame: up to 6 hours after the first dose
Population: FAS. As a standard-of-care reference arm, the "HB/APAP" arm was not intended for statistical comparisons to VX-150.
Measure: Median (Full Range); unit: minutes
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 80 | 82
minutes | 53.4 [8 to 359] | 75.9 [27 to 358]
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p = 0.3294, Regression, Cox; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.79 to 2.00]

6. Secondary Outcome: Time to First Rescue Medication After the First Dose of VX-150 Versus Placebo
Description: Time to first rescue medication was the time elapsed from the first dose of VX-150 or placebo until the participants received the first dose of rescue medication.
Time Frame: up to 48 hours after the first dose
Population: FAS. As a standard-of-care reference arm, the "HB/APAP" arm was not intended for statistical comparisons to VX-150.
Measure: Median (Full Range); unit: hours
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 80 | 82
hours | 2.7 [0.5 to 42.7] | 2.3 [0.5 to 40.2]
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p = 0.2341, Regression, Cox

7. Secondary Outcome: Percentage of Participants Using Rescue Medication After the First Dose VX-150 Versus Placebo
Time Frame: 0 to 24 hours after the first dose and 24 to 48 hours after the first dose
Population: FAS. As a standard-of-care reference arm, the "HB/APAP" arm was not intended for statistical comparisons to VX-150.
Measure: Number; unit: percentage of participants
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 80 | 82
percentage of participants
  0 to 24 hours after the first dose | 83.8 | 89.0
  24 to 48 hours after the first dose | 56.3 | 69.5
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p = 0.3358, Cochran-Mantel-Haenszel — 0 - 24 hours
Statistical Analysis 2: Comparison: VX-150 vs Placebo; Test type: Superiority; p = 0.0849, Cochran-Mantel-Haenszel — Greater than (>) 24 - 48 hours

8. Secondary Outcome: Total Rescue Medication Used After the First Dose of VX-150 Versus Placebo
Description: Total use of rescue medication was calculated as the sum of number of capsules multiplied by capsule strength at each dosing occasion of rescue medication. Rescue medication was ibuprofen (400 mg [oral] every 4 hours (q4h) as needed).
Time Frame: 0 to 24 hours after the first dose and 24 to 48 hours after the first dose
Population: FAS. As a standard-of-care reference arm, the "HB/APAP" arm was not intended for statistical comparisons to VX-150.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | VX-150 | Placebo
Number analyzed (Participants) | 80 | 82
mg
  0 to 24 hours after the first dose | 800 (341.1) | 1084.9 (478.3)
  24 to 48 hours after the first dose | 577.8 (289.9) | 786.0 (413.8)
Statistical Analysis 1: Comparison: VX-150 vs Placebo; Test type: Superiority; p = 0.0004, Wilcoxon rank-sum test — 0 - 24 hours
Statistical Analysis 2: Comparison: VX-150 vs Placebo; Test type: Superiority; p = 0.0035, Wilcoxon rank-sum test — >24 - 48 hours

9. Secondary Outcome: Maximum Observed Concentration (Cmax) of VRT- 1207355 (Active Moiety) and VRT- 1268114 (Metabolite M5)
Time Frame: Day 1 and Day 2
Population: The pharmacokinetic (PK) set included all randomized participants who received at least 1 dose of study drug. Here "Number Analyzed" signifies those participants who were evaluable at specified time points. This outcome measure is applicable to VX-150 arm only.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | VX-150
Number analyzed (Participants) | 79
microgram per milliliter (mcg/mL)
  VRT- 1207355 Day 1 | 4.95 (2.00)
  VRT- 1207355 Day 2: number analyzed (Participants) | 74
  VRT- 1207355 Day 2 | 4.92 (1.61)
  VRT- 1268114 Day 1 | 1.65 (0.779)
  VRT- 1268114 Day 2: number analyzed (Participants) | 74
  VRT- 1268114 Day 2 | 2.53 (0.797)

10. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of VRT- 1207355 and VRT- 1268114
Time Frame: Day 1 and Day 2
Population: PK set. Here "Number Analyzed" signifies those participants who were evaluable at specified time points. This outcome measure is applicable to VX-150 arm only.
Measure: Median (Full Range); unit: hours
Arm/Group | VX-150
Number analyzed (Participants) | 79
hours
  VRT- 1207355 Day 1 | 5.58 [1.08 to 12.1]
  VRT- 1207355 Day 2: number analyzed (Participants) | 74
  VRT- 1207355 Day 2 | 4.03 [0.00 to 6.25]
  VRT- 1268114 Day 1 | 8.10 [1.08 to 12.3]
  VRT- 1268114 Day 2: number analyzed (Participants) | 74
  VRT- 1268114 Day 2 | 4.03 [0.00 to 8.18]

11. Secondary Outcome: Area Under the Concentration Versus Time Curve From 0 to 12 Hours (AUC0-12h) of VRT- 1207355 and VRT- 1268114
Time Frame: Day 1 and Day 2
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: microgram*hour per milliliter (mcg*h/mL)
Arm/Group | VX-150
Number analyzed (Participants) | 79
microgram*hour per milliliter (mcg*h/mL)
  VRT- 1207355 Day 1 | 38.8 (15.9)
  VRT- 1207355 Day 2: number analyzed (Participants) | 74
  VRT- 1207355 Day 2 | 45.7 (15.5)
  VRT- 1268114 Day 1 | 12.9 (6.20)
  VRT- 1268114 Day 2: number analyzed (Participants) | 74
  VRT- 1268114 Day 2 | 25.0 (7.95)

12. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 up to Day 10
Population: The Safety Set was included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | VX-150 | HB/APAP | Placebo
Number analyzed (Participants) | 80 | 81 | 82
participants
  Participants with AEs | 25 | 30 | 29
  Participants with SAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to Day 10
Arm/Group | VX-150 | HB/APAP | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/81 | 0/82
Other Adverse Events (participants affected / at risk) | 20/80 | 22/81 | 23/82
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VX-150 (N=80) | HB/APAP (N=81) | Placebo (N=82)
Headache (Nervous system disorders) | 9 | 10 | 14
Dizziness (Nervous system disorders) | 4 | 6 | 2
Nausea (Gastrointestinal disorders) | 9 | 16 | 11
Vomiting (Gastrointestinal disorders) | 4 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT03206749/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03206749/SAP_001.pdf